CLINICAL TRIAL: NCT00951925
Title: Protocol to Obtain Bone Marrow for Research
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Christopher H. Lowrey, Professor of Medicine and of Pharmacology and Toxicology, Dartmouth-Hitchcock Medical Center
Other Study IDs: D0529
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Bone Marrow Biopsy
Keywords: diagnostic bone marrow biopsies; bone marrow harvesting for autologous BMT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 5cc of bone marrow aspirate
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No Treatment
  Interventions: Other: Bone Marrow Aspirate Draw

INTERVENTIONS:
Other: Bone Marrow Aspirate Draw — 5cc of Bone Marrow Aspirate will be drawn

SUMMARY:
Potential donors who are undergoing bone marrow biopsy or bone marrow donation as part of clinical care will be asked by the principal investigator (PI) if they might be interested in donating marrow for this research project. If they are interested, the PI will meet with the prospective donor to review the information contained in the informed consent document and to answer any questions the potential subject may have. Bone marrow aspirates of approximately 5cc will be obtained from the posterior iliac crest of subjects using standard techniques.

DETAILED DESCRIPTION:
The purpose of this study is to determine the mechanisms that regulate human globin gene expression by analyzing the function of cell signaling pathways and the expression of other related genes and their protein products in the bone marrow cells of people without blood diseases. This includes the effects of drugs and other in vitro manipulations of the cells once they are removed from donors. These assays will include, but are not limited to, determinations of DNA methylation status, histone acetylation profiles, DNAse sensitivity, transcription factor binding to DNA, levels of various proteins, messenger RNAs and miRNAs in the cells of the marrow samples. By understanding how this process occurs in people without blood diseases, we hope to to design future treatments for people with diseases such as sickle cell disease and B-thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing diagnostic bone marrow biopsies at the Norris Cotton Cancer Center of DHMC.
* Patients undergoing bone marrow harvesting for autologous bone marrow transplantation.
* Normal donors undergoing bone marrow harvesting for autologous bone marrow transplantation.
* Normal persons over the age of 17 who volunteer to undergo bone marrow aspiration.

Exclusion Criteria:

* Normal volunteers with known allergies to lidocaine (or similar analgesics)or betadine.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Patients undergoing diagnostic bone marrow biopsies at the Norris Cotton Cancer Center of Dartmouth Hitchcock Medical Center (DHMC).
  * Patients undergoing bone marrow harvesting for autologous bone marrow transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2005-06; Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Regulation of human globin gene expression | Ongoing
  The purpose of this study is to determine the mechanisms that regulate human globin gene expression by analyzing the function of cell signaling pathways and the expression of other related genes and their protein products in the bone marrow cells of people without blood diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H Lowrey, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States